CLINICAL TRIAL: NCT07394023
Title: The Effect of Mindfulness-Based Compassionate Living Practice on Stress, Pain, and Self-Efficacy in Primary Dysmenorrhea
Brief Title: The Effect of Mindfulness-Based Compassionate Living Practice on Primary Dysmenorrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Safiye AĞAPINAR ŞAHİN, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SSAHIN0002
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Mindfulness Training
Keywords: Pain; Dysmenorrhea; Mindfulness; Compassion; Stress; Self-Efficacy; Living
MeSH Terms: conditions — Pain; Dysmenorrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Session I: General Objective Group Structuring, How We Evolved - Threat, Drive, and Appeasement (Experimental): . Introduction,
  * Structuring the group process,
  * Establishing group rules and understanding their importance,
  * Informing group members about the concept of self-compassion,
  * Why Compassion? A general introduction to Evolution and Attachment Theory,
  * Threat, drive, and appeasement
  Interventions: Behavioral: Session 1: How We Evolved - Threat, Impulse, and Soothing Systems
- Session 2: Threat and Self-Compassion (Experimental): * A "breath break with kindness" is practiced. • "Building a compassionate relationship with resilience" and "kindness meditation: a benevolent" practices are made. • "A hand on your heart" and "a compassionate comrade" practices are made.
  Interventions: Behavioral: Session 2: Threat and Self-Compassion
- Session 3: Unraveling the Knots of Desire and Patterns Agenda (Experimental): * Talk about homework. • A "breath break with kindness" is practiced.
  * Establishing a compassionate relationship with desire", "guided meditation to discover the inner pattern", "courtesy meditation: a good friend" practices are made.
  Interventions: Behavioral: Session 3: Unraveling the Knots of Desire and Patterns
- Session 4: Internalizing compassion (Experimental): * "Pretend-to-pretend" practice is made for participants to observe themselves. • In addition to the previous practices, the practice of "internalizing compassion" is made in order to increase their expanded mindfulness.
  • Courtesy meditation: a neutral person", "kindness towards your body", which is based on mindfulness practices and increases body awareness and mindful movement, is carried out. During the day, they will be informed that they should do the "walking with kindness" practice on their own
  Interventions: Behavioral: Session 4: Internalizing compassion
- Session 5: Me and others - Expanding the circle (Experimental): * A "compassionate letter" application is made by asking participants to think about a situation they encountered recently or some time ago and is still causing distress. It is explained that they can gain insight with this application. • "Courtesy meditation: the 'difficult' person", "compassion and breathing: yourself" and "compassionate breathing: others" practices are made
  Interventions: Behavioral: Session 5: Me and others - Expanding the circle
- Session 6: Growing happiness (Experimental): * "Revisiting the good" practice is carried out to define the five sense organs for the participants. • "Forgiveness", "Asking for forgiveness", "forgiving others", "gratitude" practices are carried out. • The practice is expanded as "kindness meditation: groups and all beings".
  Interventions: Behavioral: Session 6: Growing happiness
- Session 7: Weaving Wisdom and Compassion into Daily Life (Experimental): * Participants are made to choose a day in their life and allow a few minutes to pause in a mindful way.
  • "A breather for wise and compassionate action", "calmness meditation" and "joy sharing meditation" practices are carried out.
  Interventions: Behavioral: Session 7: Weaving Wisdom and Compassion into Daily Life
- Session 8: Living with the Heart (Experimental): * The participants are told about the applications that they can apply for, where they need help to develop compassion towards self-healing skills, and the whole training is evaluated. • The "river of life" application, which evaluates mindfulness in depth, is carried out.
  • An overall summary of the 8-session study is made and feedback is received.
  Interventions: Behavioral: Session 8: Living with the Heart

INTERVENTIONS:
Behavioral: Session 1: How We Evolved - Threat, Impulse, and Soothing Systems — The practice of "Breath break with kindness" will be applied for 5 minutes. Afterwards, 15 minutes of information on threats, impulses and soothing systems, "A safe place" application for 11 minutes, "Courtesy meditation" for 10 minutes. After each application, 10 minutes of feedback will be received from the participants.
  Arms: Session I: General Objective Group Structuring, How We Evolved - Threat, Drive, and Appeasement
Behavioral: Session 2: Threat and Self-Compassion — The practice of "breathing with kindness" will be done for 7 minutes. The practice of "Building a compassionate relationship with resilience" will be held for 12 minutes, and the practice of "Kindness meditation: a benevolent" will take place for 11 minutes. "A hand over your heart" application will be made for 3 minutes and "A compassionate comrade" application will be done for 10 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 2: Threat and Self-Compassion
Behavioral: Session 3: Unraveling the Knots of Desire and Patterns — The practice of "breathing with kindness" will be done for 7 minutes. "Building a compassionate relationship with desire" 12 minutes, "Guided meditation to discover the inner pattern" 10 minutes and "Courtesy meditation: a good friend" 11 minutes. Except for the "breath break with kindness" application, 3 minutes of feedback will be received from the participants after each application
  Arms: Session 3: Unraveling the Knots of Desire and Patterns Agenda
Behavioral: Session 4: Internalizing compassion — The "pretend-to-be" practice for the participants to observe themselves will be made for 10 minutes. The practice of "internalizing compassion" will be done for 7 minutes, "kindness meditation: a neutral person" practice for 10 minutes, and "kindness towards your body" for 10 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 4: Internalizing compassion
Behavioral: Session 5: Me and others - Expanding the circle — The "a compassionate letter" practice with the participants will continue for 15 minutes. "meditation: the 'difficult' person" 8 minutes, "compassion and breathing: yourself" 10 minutes and "compassionate breathing: others" 7 minutes. A "compassionate break" application is performed for 7 minutes.
  Arms: Session 5: Me and others - Expanding the circle
Behavioral: Session 6: Growing happiness — The practice of "Revisiting the good" is carried out for 10 minutes with the participants. "Forgive yourself", "wish for forgiveness", "forgive others", "gratitude" practices will be held for 5 minutes each and will take 20 minutes in total. "Courtesy meditation: groups and all beings" will be practiced for 10 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 6: Growing happiness
Behavioral: Session 7: Weaving Wisdom and Compassion into Daily Life — Participants will be given 10 minutes to choose a day in their life and allow a few minutes to pause mindfully. The practice of "a breather for wise and compassionate action" is 10 minutes, the practice of "calmness meditation" is 8 minutes, and the practice of "sharing the joy meditation" is 8 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 7: Weaving Wisdom and Compassion into Daily Life
Behavioral: Session 8: Living with the Heart — The participants are told about the applications they can apply for, where they need help to develop compassion towards self-healing skills, and the entire training will be evaluated for 20 minutes. The "river of life" application is carried out for 20 minutes. 10 minutes of feedback will be received after the application.
  Arms: Session 8: Living with the Heart

SUMMARY:
This study aims to evaluate the effects of "Mindfulness-Based Self-Compassion Training" given to students with Primary Dysmenorrhea on Stress, Pain, and Self-Efficacy. The research will be conducted at Atatürk University Faculty of Health Sciences between October 2025 and October 2026. The study was conducted with individuals who met the inclusion criteria and agreed to participate. Data were collected using a Sociodemographic Information Form, Visual Analog Scale (VAS), Perceived Stress Scale (PSS), Self-Efficacy Scale (SES), Self-Compassion Scale Short Form (SCS-S), and Mindfulness Scale (MSS). After collecting pre-test data, students with PMS in the experimental group received 8 sessions of Mindfulness-Based Self-Compassion training. The first two sessions were conducted face-to-face, and the remaining sessions were conducted online. No intervention was applied to the control group. The sample size of the study was calculated using the GPower computer program. A power analysis performed at α=0.05 yielded an effect size of 150,153 (d=0.8), achieving 90% power. Therefore, it was calculated that the sample should include at least 68 participants. This research is being conducted with 68 participants.

DETAILED DESCRIPTION:
Data was collected through face-to-face interviews by the researcher. Women meeting the inclusion criteria (women experiencing Primary Dysmenorrhea, those scoring 45 or higher on the Visual Analog Scale) were included in the study. Pre-test assessment tools were administered to the participants. The experimental group received 40 minutes of Mindfulness-Based SelfCompassion training once a week for 8 weeks. The control group received no intervention. Post-test data will be collected after the training sessions.

ELIGIBILITY:
Inclusion Criteria:

* Students with regular menstrual periods (lasting 3-8 days, with a menstrual cycle range of 21-35 days),
* Students with dysmenorrhea pain intensity of 45 mm or more according to the Visual Analog Scale (VAS).

Exclusion Criteria:

* Students diagnosed with secondary dysmenorrhea (endometriosis, ovarian cyst/tumor, pelvic infectious disease, myoma, uterine polyps, uterine adhesions, infection, etc.),
* Students using oral contraceptives,
* Students with compromised tissue integrity in the abdominal area,
* Students with any chronic or mental illness.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 68 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Demographic Information Form: | up to 1 day
  This form consists of 14 questions prepared by the researcher in accordance with the relevant literature. It includes questions about students' demographic information (age, department, class, marital status, and place of residence) and characteristics of their menstrual cycle (age of menarche, duration of bleeding and pain, etc.).

SECONDARY OUTCOMES:
Visual Analog Scale (VAS): | up to 1 day
  VAS is used to measure the pain perceived by a person. Between a 10 cm (100 mm) section of the scale, where one end is marked with no pain (zero) and the other end with the most severe pain (10), the individual can indicate their pain by drawing a line, placing a dot, or marking it. The distance from the point where there is no pain to the point marked by the individual is measured in centimeters, and the resulting value indicates the severity of the individual's pain. On the VAS scale, 0-44 mm indicates mild pain, 45-74 mm indicates moderate pain, and 75-100 mm indicates severe pain (Tulunay and Tulunay, 2000).

OTHER OUTCOMES:
Perceived Stress Scale (PSS): | up to 1 day
  Developed by Cohen, Kamarck, and Mermelste in 1983, was used to determine the perceived stress level of the participants (Appendix-7).
  The Cronbach alpha value was found to be 0.86 in the reliability study of the scale.
  The adaptation of the scale into Turkish was done by Bilge, Öğce, Genç, and Oran (2007), and the Cronbach alpha value was found to be 0.82 in the reliability study.
  The scale includes some situations containing the feelings and thoughts that individuals may have experienced during the past month. Individuals indicated how often they experienced each situation in the past month.
  The scale, prepared with a five-point Likert type (0 never, 4 very often), has three items that are reversed (items 4, 5, 6) and five items that are direct (items 1, 2, 3, 7, 8). A total score between 0 and 32 is obtained from the scale. The scale has two subscales: perceived stress (items 1, 2, 3, 7, 8) and perceived coping (items 4, 5, 6). The scale is evaluat
Short Form of Self-Compassion Scale (SSS-C) | up to 1 day
  The Turkish validity and reliability of the scale developed by Neff (2003) was made by Yıldırım and Sarı in 2018.
  The scale was confirmed to have a structure consisting of 11 items, a single dimension and two complementary components (positive component and negative component). The internal consistency coefficient of the scale was calculated as .75. Gerber (2021) used the scale developed by Neff (2003) and a professional caregiver working in the intensive care and rehabilitation units of a hospital, and reported that self-compassion is a factor associated with reducing the level of burnout in individuals. It is recommended to be used in studies where a total score will be made to measure self-compassion.
Mindfulness Awareness Scale (MAS): | up to 1 day
  Developed by Brown and Ryan (2003) to assess individuals' level of mindfulness. Its Turkish validity and reliability were established by Özyeşil et al. (2011). The scale is a unidimensional, six-point Likert-type scale consisting of 15 questions. The Cronbach's alpha coefficient of the scale was determined to be 0.80. The minimum and maximum scores individuals can obtain on the scale range from 15 to 90. Higher scores indicate a higher level of mindfulness.

IPD SHARING:
Plan to Share IPD: No